CLINICAL TRIAL: NCT03795792
Title: Efficacy of Oral Curcumin Administration on Metabolic Syndrome Remission.
Brief Title: Oral Curcumin Administration to Remit Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Fernando Guerrero Romero MD, Head of the research unit, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2017-785-132
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Study groups:
  Intervention group: curcumin 1.2 g / black pepper 10 mg a day for 3 months, plus recommendations to decrease calories intake and do exercise.
  Control group: hydrolyzed collagen 1.2 g / black pepper 10 mg a day for 3 months, plus recommendations to decrease calories intake and do exercise.
Who Masked: Participant, Care Provider
Masking Description: Neither the patient nor the treating doctor will know the study group the participant was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin (Experimental): Curcumin 1.2 g / black pepper 10 mg a day for 3 months, plus recommendations to decrease calories intake and do exercise.
  Interventions: Dietary Supplement: Curcumin
- Hydrollased collagen (Placebo Comparator): Hydrolyzed collagen 1.2 g / black pepper 10 mg a day for 3 months, plus recommendations to decrease calories intake and do exercise.
  Interventions: Dietary Supplement: Hydrolyzed collagen

INTERVENTIONS:
Dietary Supplement: Curcumin — Will be provided in capsules
  Other Names: Turmeric
  Arms: Curcumin
Dietary Supplement: Hydrolyzed collagen — Will be provided in capsules.
  Arms: Hydrollased collagen

SUMMARY:
The metabolic syndrome consists of a set of risk factors that increases the probability to develop heart diseases and type 2 diabetes, two of the principal chronic diseases that affect Mexican population. The curcumin is a compound that is extracted from the root of a plant called Cúrcuma longa. There exists information that curcumin helps to diminish weight and the levels of blood glucose and blood fats. The hypothesis of this study is: that curcumin administration combined with diet and exercise remits the metabolic syndrome.

DETAILED DESCRIPTION:
Objective: The aim of this study is to determinate the efficacy of oral administration of curcumin in the remission of metabolic syndrome.

Design: clinical trial, randomized, double blind, placebo controlled.

Study population: Men and women from 20 to 55 years old with metabolic syndrome according to the ATP III criteria, will be included.

Study groups: intervention and control group.

Sample size: It was calculated using a statistical power of 80%, an alpha value of 0.05. A 50% of the difference in the mean of remission of metabolic syndrome between control group and intervention groups was considered. The estimated sample size was 220 subjects for each group.

Process: All eligible participants according to inclusion and exclusion criteria, will be randomized to one of the study groups.

The intervention group will receive a total dose of curcumin 1.2 g / black pepper 10 mg a day; and control group will receive a total dose of hydrolyzed collagen 1.2 g / black pepper 10 mg a day; plus dietary and exercise recommendations for both groups during three months.

The blood concentrations of glucose, triglycerides, and HDL cholesterol will be measured, as well as the abdominal perimeter and blood pressure, at baseline conditions, at one month and three months after treatment.

Statistical analysis: Numerical values will be expressed as mean ± standard deviation; categorical variables will be expressed as proportions. Differences between the groups were estimated by unpaired Student t test for numerical variables (Mann-Whitney U test for skewed data) or Chi-square and Fisher´s exact test for categorical variables. Intragroup differences were estimated by paired Student t-test.

ELIGIBILITY:
Inclusion Criteria:

* Women and men.
* 20 to 55 years old.
* Diagnosis of metabolic syndrome according to the ATP III criteria.
* Informed consent of the participant.

Exclusion Criteria:

* Diabetes or hypoglycaemic therapy.
* High blood pressure o anti-hypertensive treatments.
* Hypertriglyceridemia (>400 g/dL) or lipid lowering treatment.
* Neoplasia disease.
* Thyroid disease
* Syndrome of polycystic ovary.
* Pregnancy or lactation.
* Smoking.
* Anti-inflammatory medicines in the last two months.
* Food supplements in the last two months.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Remission of metabolic syndrome. | Three months.
  Presence of two or less metabolic syndrome criteria, according to the ATP III criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Guerrero, PhD, Principal Investigator — Instituto Mexicano del Seguro Social; Luis Simental, PhD, Study Chair — Instituto Mexicano del Seguro Social; Gerardo Martínez, PhD, Study Chair — Instituto Mexicano del Seguro Social; Claudia Gamboa, PhD, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Biomedical Research Unit. IMSS. Durango, Durango, Durango, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azhar Y, Parmar A, Miller CN, Samuels JS, Rayalam S. Phytochemicals as novel agents for the induction of browning in white adipose tissue. Nutr Metab (Lond). 2016 Dec 3;13:89. doi: 10.1186/s12986-016-0150-6. eCollection 2016. PMID 27980598
- [Background] Cabrera-Rode E, Stusser B, Calix W, Orlandi N, Rodriguez J, Cubas-Duenas I, Echevarria R, Alvarez A. [Diagnostic concordance between seven definitions of metabolic syndrome in overweight and obese adults]. Rev Peru Med Exp Salud Publica. 2017 Jan-Mar;34(1):19-27. doi: 10.17843/rpmesp.2017.341.2763. Spanish. PMID 28538842
- [Background] Di Pierro F, Bressan A, Ranaldi D, Rapacioli G, Giacomelli L, Bertuccioli A. Potential role of bioavailable curcumin in weight loss and omental adipose tissue decrease: preliminary data of a randomized, controlled trial in overweight people with metabolic syndrome. Preliminary study. Eur Rev Med Pharmacol Sci. 2015 Nov;19(21):4195-202. PMID 26592847
- [Background] Jimenez-Osorio AS, Monroy A, Alavez S. Curcumin and insulin resistance-Molecular targets and clinical evidences. Biofactors. 2016 Nov 12;42(6):561-580. doi: 10.1002/biof.1302. Epub 2016 Jun 21. PMID 27325504
- [Background] Kim M, Kim Y. Hypocholesterolemic effects of curcumin via up-regulation of cholesterol 7a-hydroxylase in rats fed a high fat diet. Nutr Res Pract. 2010 Jun;4(3):191-5. doi: 10.4162/nrp.2010.4.3.191. Epub 2010 Jun 28. PMID 20607063
- [Background] Metzler M, Pfeiffer E, Schulz SI, Dempe JS. Curcumin uptake and metabolism. Biofactors. 2013 Jan-Feb;39(1):14-20. doi: 10.1002/biof.1042. Epub 2012 Sep 20. PMID 22996406
- [Background] Mohammadi A, Sahebkar A, Iranshahi M, Amini M, Khojasteh R, Ghayour-Mobarhan M, Ferns GA. Effects of supplementation with curcuminoids on dyslipidemia in obese patients: a randomized crossover trial. Phytother Res. 2013 Mar;27(3):374-9. doi: 10.1002/ptr.4715. Epub 2012 May 21. PMID 22610853
- [Background] Na LX, Yan BL, Jiang S, Cui HL, Li Y, Sun CH. Curcuminoids Target Decreasing Serum Adipocyte-fatty Acid Binding Protein Levels in Their Glucose-lowering Effect in Patients with Type 2 Diabetes. Biomed Environ Sci. 2014 Nov;27(11):902-6. doi: 10.3967/bes2014.127. PMID 25374024
- [Background] Na LX, Li Y, Pan HZ, Zhou XL, Sun DJ, Meng M, Li XX, Sun CH. Curcuminoids exert glucose-lowering effect in type 2 diabetes by decreasing serum free fatty acids: a double-blind, placebo-controlled trial. Mol Nutr Food Res. 2013 Sep;57(9):1569-77. doi: 10.1002/mnfr.201200131. Epub 2012 Aug 29. PMID 22930403
- [Background] Neyrinck AM, Alligier M, Memvanga PB, Nevraumont E, Larondelle Y, Preat V, Cani PD, Delzenne NM. Curcuma longa extract associated with white pepper lessens high fat diet-induced inflammation in subcutaneous adipose tissue. PLoS One. 2013 Nov 19;8(11):e81252. doi: 10.1371/journal.pone.0081252. eCollection 2013. PMID 24260564
- [Background] Rahimi HR, Mohammadpour AH, Dastani M, Jaafari MR, Abnous K, Ghayour Mobarhan M, Kazemi Oskuee R. The effect of nano-curcumin on HbA1c, fasting blood glucose, and lipid profile in diabetic subjects: a randomized clinical trial. Avicenna J Phytomed. 2016 Sep-Oct;6(5):567-577. PMID 27761427
- [Background] Kowluru RA, Kanwar M. Effects of curcumin on retinal oxidative stress and inflammation in diabetes. Nutr Metab (Lond). 2007 Apr 16;4:8. doi: 10.1186/1743-7075-4-8. PMID 17437639
- [Background] Rochlani Y, Pothineni NV, Kovelamudi S, Mehta JL. Metabolic syndrome: pathophysiology, management, and modulation by natural compounds. Ther Adv Cardiovasc Dis. 2017 Aug;11(8):215-225. doi: 10.1177/1753944717711379. Epub 2017 Jun 22. PMID 28639538
- [Background] Shao W, Yu Z, Chiang Y, Yang Y, Chai T, Foltz W, Lu H, Fantus IG, Jin T. Curcumin prevents high fat diet induced insulin resistance and obesity via attenuating lipogenesis in liver and inflammatory pathway in adipocytes. PLoS One. 2012;7(1):e28784. doi: 10.1371/journal.pone.0028784. Epub 2012 Jan 9. PMID 22253696
- [Background] Shen L, Ji HF. The pharmacology of curcumin: is it the degradation products? Trends Mol Med. 2012 Mar;18(3):138-44. doi: 10.1016/j.molmed.2012.01.004. Epub 2012 Mar 1. PMID 22386732
- [Background] Shin SK, Ha TY, McGregor RA, Choi MS. Long-term curcumin administration protects against atherosclerosis via hepatic regulation of lipoprotein cholesterol metabolism. Mol Nutr Food Res. 2011 Dec;55(12):1829-40. doi: 10.1002/mnfr.201100440. Epub 2011 Nov 7. PMID 22058071
- [Background] Yang YS, Su YF, Yang HW, Lee YH, Chou JI, Ueng KC. Lipid-lowering effects of curcumin in patients with metabolic syndrome: a randomized, double-blind, placebo-controlled trial. Phytother Res. 2014 Dec;28(12):1770-7. doi: 10.1002/ptr.5197. Epub 2014 Aug 6. PMID 25131839